CLINICAL TRIAL: NCT05730374
Title: Effect of Benson's Relaxation Technique Versus Music Therapy on Physiological Parameters and Stress of Children With Thalassemia During Blood Transfusion
Brief Title: Benson's Relaxation Technique, Music Therapy for Children With Thalassemia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Alexandria University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: BRT
Record Dates: First submitted 2023-01-24; First posted 2023-02-15 (Actual); Last update posted 2023-07-20 (Actual); Status verified 2023-01

CONDITIONS: Thalassemia in Children
Keywords: Benson's Relaxation; Music Therapy; Stress; Thalassemia
MeSH Terms: conditions — Thalassemia | interventions — Music Therapy

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (No Intervention): children with thalassemia will receive only routine care of hospital during blood transfusion.
- Benson's Relaxation Group (Experimental): children with thalassemia will receive Benson's relaxation intervention beside routine care of hospital during blood transfusion
  Interventions: Behavioral: Benson's Relaxation technique
- Music Therapy Group (Experimental): children with thalassemia will receive music therapy intervention beside routine care of hospital during blood transfusion.
  Interventions: Behavioral: Music therapy

INTERVENTIONS:
Behavioral: Benson's Relaxation technique — Each child in the study group had an individual interview with researchers, who demonstrated the Benson relaxation technique while teaching them. The child was then asked to demonstrate it. sit quietly in a comfortable position in separate room., close eyes, deeply relax all muscles, beginning at the feet and progressing up to the face and breathe through nose. Become aware of breathing pattern. As breathes out, say the word one silently to child. For example, breathe in, and then out, say one, in and out, and repeat one. Breathe easily and naturally. It is Continue for 10 minutes and repeated two times.
  Arms: Benson's Relaxation Group
Behavioral: Music therapy — * The child lessen to a Mozart's music, which is played before and throughout the blood transfusion procedure. Ambient noise can be reduced by using headphones. As a result, it is easier to see how the intervention has succeeded.
  * This intervention was done using an MP3 player during the blood transfusion procedure and immediately following the completion of the intervention to prevent the transmission of infections headphones were cleaned with disinfectant after each -use.
  Arms: Music Therapy Group

SUMMARY:
The aim of the present study is to determine the effect of Benson's relaxation technique versus music therapy on physiological parameters and stress of children with thalassemia during blood transfusion.

DETAILED DESCRIPTION:
Thalassemia is the most common hematological disease in Egypt and the world that is transmitted by parents to their children and has no definitive cure. It means a group of hereditary blood diseases caused by defects haemoglobin (Hb) synthesis that results from an alteration in the gene responsible for producing globin chains leading to alteration in the rate of its production .

Generally in worldwide, There are about 300 million thalassemia patients, 55 million of whom live in Southeast Asia . In Egypt, beta-Thalassemia represents a major public health problem. It is reported that the carrier rate is between 9 to 10% of the population. It has been estimated that one thousand children out of 1.5 million live births are born each year suffering from thalassemia. In spite of optimal treatment being available, only a few children can afford it. Unfortunately, most children suffer from complications of blood transfusions, mainly transfusion transmitted viral infections and iron overload. Prevention by carrier detection and prenatal diagnosis is needed in populations with high incidence of the disease, such as Egypt.

The most severe form is the β-thalassemia major, which is characterized by a severe microcytic, hypochromic anemia (Cooley's anemia), whose symptoms appear usually within the first 2 years of life due to iron overload. Chronic iron overload can occur in children with beta-thalassemia as may need blood transfusions throughout their life. Iron overload can lead to growth retardation, pallor, poor appetite, and often jaundice; as well as hinder sexual development during the adolescent period and dysfunction of organs, such as heart, pancreas, and endocrine glands.

When the storage capacity of the body is exceeded, iron remains in free form. The formation of hydroxyl free radicals can be catalyzed by this free iron, leading to damage of cell membranes and protein denaturation. Ultimately, tissue damage occurs which can lead to significant levels of morbidity and mortality. Iron chelation helps prevent complications of iron overload due to repeated blood transfusion. Indeed, the most common complication of beta-thalassemia that leads to death is organ failure, in children taking regular blood transfusions and no appropriate iron chelation. Elevated liver iron concentrations (LICs) and serum ferritin levels can manifest within 1-2 years of starting regular blood transfusions. Children with thalassemia whose serum ferritin level is more than 2500 ng/mL or LIC value is more than 15 mg Fe/kg dry weight are at high risk of development of cardiac diseases such as cardiomyopathy.

Significant advances in treatment modalities and improved clinical management have led to a substantially higher life expectancy of these children. Children with thalassemia major have good survival but little is known about their psychological status. children are less able to voice their concerns and are more vulnerable than adults.

Today, with the help of existing therapies and the use of new drugs to improve iron overload control and timely initiation of treatment, the disease has become a chronic disease and life expectancy in these children has increased. However, repeated blood transfusions and long-term use of iron-chelating drugs affect other aspects of these children' lives and significantly affect their general health, mental health, and quality of life, and their families.

Thalassemia can cause different physiological, emotional, social, financial and behavioral problems that affect the life of both patients and their families, its effects are stronger particularly during school age and adolescence. It can greatly affect the sense of autonomy and mental health. Children with thalassemia major experience a lot of stress throughout their lives which constituted 18.8 %. Successive blood tests for fatigue, fatigue from successive blood transfusions, and subcutaneous injections of iron chelators, in addition to the body, irritate the souls of these patients. So much so that most of these patients also have mental disorders. It was described the fear and anxiety caused by injections in these children as the most difficult aspect of their illness.

Physiological changes occur when a person is threatened with illness, trauma, or stress. The physiological response to the stressor in the cardiovascular system increases blood pressure, changes the number of pulses and respiration, increases oxygen saturation, and increases the risk of arrhythmias. Therefore, it is very important to find an effective solution that is also cost-effective for clinical use.

Stress can be defined as any uncomfortable or agonizing emotional experience associated with changes in behavior as well as biochemical and physiological changes or in simple words we can say it is a feeling of being worried or overwhelmed. It can affect anyone regardless of age or gender of person and result in both physical as well as psychological health issues. Stress among children with thalassemia can be attributed to number of reasons like frequent treatment procedures and hospital visits, decreased life expectancy, expected complications from disease or treatment procedures and the monetary burden on parents. Also, the long painful treatment sessions such as to remove iron as iron overload being a complication of frequent blood transfusions, and an eight hour long painful procedure when injecting chelators by chelation pump is carried out, adding to the stress factors.

Unlike pharmacological treatments, complementary therapies in addition to cost effective, have no serious side effects or drug interactions, they are easy to perform, and well accepted by the patient. It is important to pay attention to additional therapies in the sense that can be performed by nurses without the need for a doctor's prescription, as well as to pave the way for nurses to gain professional independence.

Relaxation is one of the best complementary treatment strategies to decrease stress and mental disorders of the patients in order to improve their physical, psychological, and social functions. Moreover, relaxation increases the secretion of endorphins or analgesic hormone, but reduces the secretion of adrenaline hormone. In the present study, relaxation refers to one of the methods of concentration which is introduced due to its ease of learning and teaching. It was carried out in 4 stages: providing a relaxed environment, being in an appropriate physical position, concentration and creation of an inactive state. Creation of a calm environment, reduce muscle tension and focus by focusing on one word, increasing a person's attention, reducing the number of breaths and lactate in the blood can be occurred in Benson muscle relaxation due to lack of muscle stiffness, number of breaths, pulse and blood pressure are not increased and cardiac output is not increased.

So Benson relaxation therapy, as well as other relaxation techniques, that may cause a decrease in physical and psychological stress, which conceptually can decrease epinephrine, decrease cortisol, decrease glucagon and decrease thyroid hormone. All of these have a positive effect on reducing stress levels. Reduction in stress levels and the attainment of a relaxed condition in patients have positive effect on reducing stress levels. Therefore, various efforts were made to make patients comfortable and remain relaxed.

In addition to the Benson relaxation techniques described above, music therapy is another non-pharmacological methods that is believed to provide a relaxing effect on the patient and it considered to help reduce and even overcome psychological disorders and discomforts such as anxiety, stress, depression, and so on. Music therapy can be defined as the prescribed and organized use of music or its activities to change the maladaptive state in order to help clients achieve therapeutic goals. Music reduces stress by distracting and reducing a person's focus on stressful stimuli. Physicians can use it to reduce stress in children undergoing treatment or those with the possibility of further treatment. Due to the fact that therapeutic music has no side effects, in addition to this, it is easy, cheap, and safe and can be accepted by the client. Numerous studies have examined the effect of music therapy on reducing stress levels and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* preschool stage

Exclusion Criteria:

* Free from any neurological disorders.
* Free from major congenital malformations.

Ages: 3 Years to 6 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 120 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-04-30 (Actual)

PRIMARY OUTCOMES:
Tool I: Characteristics of Children with Thalassemia and Their Physiological Parameters Assessment Sheet: | children's characteristics will be assessed initially, pre-procedure. physiological parameters of children will be assessed as the following; • "Baseline, pre-blood transfusion procedure" • "During the blood transfusion procedure" • "Immediately after th
  This tool was developed by the researcher after reviewing the literature to assess the characteristics of children with thalassemia and their parameters. It includes two parts:Part One: children's characteristics: age, sex, and medical history. level of education, place of residence, Part Two: children's physiological parameters: respiratory rate, heart rate, and O2 saturation.

SECONDARY OUTCOMES:
Tool II: Observational Scale of Behavioral Distress: | Children's behavioral reactions to stress will be assessed as the following;• "Baseline, pre-blood transfusion procedure" • "During the blood transfusion procedure" • "Immediately after the blood transfusion procedure"
  This tool will be modified in this study to assess children's behavioral reactions to stress during a blood transfusion. It consists of an eleven-item revision of the Procedure Behavior Rating Scale, which depend on the Self-Report Measures of Fear. Children will be asked to rate "how scared" could be felt about their planned blood transfusion. Three faces were employed on a "face" scale, with the "happy" face denoting "not at all scared" and scored with 1, and the "sad" face denoting "very scared", and scored with 3. Total score of tool was ranged between 11 to 33. Children' perceived stress level will categorized as follows:
  * Mild level of stress → 11-17.
  * Moderate level of stress →18-25.
  * Severe level of stress →26-33.

CONTACTS AND LOCATIONS:
Locations (1):
- the Hematology Out-Patient Clinic of the Children's University Hospital at El-Shatby, Alexandria, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] El-said S, Darwish A, Abdelrahman D. Stress, anxiety and depression among adolescents suffering from thalassemia. Port Said Scientific Journal of Nursing, 2021;8(3): 149-61. DOI: 10.21608/PSSJN.2021.78945.1112 https://pssjn.journals.ekb.eg/article_212190.html
- [Background] El-Shanshory MR, Sherief LM, Hassab HM, Ragab SM, Yahia S, Mansour AK, Ahmed AS, Abdou SH, Helmy AM, Watany MM, Gad ALllah AM, Guindy MA, Mourad ZI, Soliman MA, El-Farahaty RM, El-Dahtory F, Darwish A, Elmabood SA, Kabbash IA, Saied SM. Prevalence of iron deficiency anemia and beta thalassemia carriers among relatives of beta thalassemia patients in Nile Delta region, Egypt: a multicenter study. J Egypt Public Health Assoc. 2021 Oct 11;96(1):27. doi: 10.1186/s42506-021-00088-9. PMID 34633587
- [Background] Hisam A, Khan NUS, Tariq NA, Irfan H, Arif B, Noor M. Perceived stress and monetary burden among thalassemia patients and their caregivers. Pak J Med Sci. 2018 Jul-Aug;34(4):901-906. doi: 10.12669/pjms.344.15420. PMID 30190750
- [Background] Jajhara I, Choudhary G, Singh J, Chachan V, Kumar A. A study on quality of life among thalassemic children aged 8 to 18 years. Int J Contemp Pediatr 2021; 8: 1667-74. DOI: https://dx.doi.org/10.18203/2349-3291.ijcp20213727.
- [Background] Kaviani M, Bahoosh N, Azima S, Asadi N, Sharif F, Sayadi M. The effect of relaxation on blood sugar and blood pressure changes of women with gestational diabetes: a randomized control trial. Iranian journal of diabetes and obesity, 2014; 6(1): 14-22
- [Background] Panigrahi M, Swain TR, Jena RK, Panigrahi A, Debta N. Effectiveness of Deferasirox in Pediatric Thalassemia Patients: Experience from a Tertiary Care Hospital of Odisha. Indian J Pharmacol. 2020 May-Jun;52(3):172-178. doi: 10.4103/ijp.IJP_68_18. Epub 2020 Aug 4. PMID 32873999
- [Background] Seifi L, Najafi Ghezeljeh T, Haghani H. The effects of benson relaxation technique and nature sound's on anxiety in patients with heart failure. Nurs Midwifery J. 2017; 15 (2):147-158. http://unmf.umsu.ac.ir/article-1-3036-en.html
- [Background] Sheikhi, A. R., Naderifar, M., Abdullahi M. A, Mastalizadeh, H., Sheikhi, H. R.The Effect of Music Therapy on the Anxiety Level of Children with Thalassemia Major under Blood Transfusion. Arch Pharma Pract 2020; 11(S4):66-9. https://www.researchgate.net/publication/348592642
- [Background] Foley V. Clinical Measurement. In: Delves -Yates, C. (Ed.) Essentials of Nursing Practice. London: Sage Co., 2015; 349-378.
- [Background] Packyanathan JS, Lakshmanan R, Jayashri P. Effect of music therapy on anxiety levels on patient undergoing dental extractions. J Family Med Prim Care. 2019 Dec 10;8(12):3854-3860. doi: 10.4103/jfmpc.jfmpc_789_19. eCollection 2019 Dec. PMID 31879625
- [Background] Poorolajal J. Effect of Benson relaxation technique on the preoperative anxiety and hemodynamic status: A single blind randomized clinical trial, 2017; 17 (1): 33 - 38
- [Background] Abd Elgwad F. Relaxation Therapy, Preeclampsia Effect of Benson's Relaxation Therapy on Stress and Physiological Parameters among Women with Preeclampsia. ASNJ, 2021;.23 (1) :63-74.
- [Background] Ali Mansouri. Evaluation of the effect of foot reflexology massage on vital signs and anxiety after blood transfusions in children with thalassemia. Bali Medical Journal, 2017; 6(3) : 623-629 ISSN.2089-1180, E-ISSN.2302-2914444444
- [Background] Salehipour S , Ghaljeh M .The Effect of Benson RelaxationTechnique on Anxiety and Aggression in Patients with Thalassemia Major: a Clinical Trial Study. P J M H S, 2021; 15( 3): 753.
- [Background] Wu PY, Huang ML, Lee WP, Wang C, Shih WM. Effects of music listening on anxiety and physiological responses in patients undergoing awake craniotomy. Complement Ther Med. 2017 Jun;32:56-60. doi: 10.1016/j.ctim.2017.03.007. Epub 2017 Mar 31. PMID 28619305
- [Background] Salkhordeh H, Sabet B, mahboobi M, Babajani S. The Effect of Music Therapy on Preoperational Anxiety and Pain in Waiting Room. Paramedical Sciences and Military Health. 2017; 12 (2) :55-62
- [Background] Najafi S S. The Effect of Music Therapy on the Level of Anxiety and vital Signs in Patients undergoing trans-esophageal Echocardiography . JAP. 2018; 9 (1) :1-11
- [Background] Ghanbari N, The Effect of Music Therapy on Pain and Anxiety of Children Diagnosed with Leukemia during P 19271 - 19286 Received 25 April 2021; Accepted 08 May 2021. 19271 http://annalsofrscb.ro
- [Background] Daneshpajooh L, Najafi Ghezeljeh T, Haghani H. Comparison of the effects of inhalation aromatherapy using Damask Rose aroma and the Benson relaxation technique in burn patients: A randomized clinical trial. Burns. 2019 Aug;45(5):1205-1214. doi: 10.1016/j.burns.2019.03.001. Epub 2019 Apr 2. PMID 30948278
- [Background] Kurniasari AN, Kustanti A, Harmilah H. The effect Benson relaxation technique with anxiety in hemodialysis patients in Yogyakarta. Indonesian J Nurs Pract 2016;1:40-7.
- [Background] Mosher CE, Jaynes HA, Hanna N, Ostroff JS. Distressed family caregivers of lung cancer patients: an examination of psychosocial and practical challenges. Support Care Cancer. 2013 Feb;21(2):431-7. doi: 10.1007/s00520-012-1532-6. Epub 2012 Jul 14. PMID 22797839
- [Background] Abarghoee SN, Mardani A, Baha R, Aghdam NF, Khajeh M, Eskandari F, Vaismoradi M. Effects of Benson Relaxation Technique and Music Therapy on the Anxiety of Primiparous Women Prior to Cesarean Section: A Randomized Controlled Trial. Anesthesiol Res Pract. 2022 Dec 23;2022:9986587. doi: 10.1155/2022/9986587. eCollection 2022. PMID 36589598
- [Background] Buckley SJ. Executive Summary of Hormonal Physiology of Childbearing: Evidence and Implications for Women, Babies, and Maternity Care. J Perinat Educ. 2015;24(3):145-53. doi: 10.1891/1058-1243.24.3.145. PMID 26834435
- [Background] Najafighazaljeh S. Comparison of Benson's Muscle Relaxation and Voice of Nature on Anxiety in Patients with Heart Failure: A Randomized Clinical Trial with Control Group. Urmia Nur and Mid J, 2017;15(2): 147
- [Background] Cahyat Y, Rosdiana I, Elengoe A, Podder S. Effect of Benson Relaxation and Aromatherapy on Blood Glucose Levels in Patients With Type II Diabetes Mellitus. Mal J Med Health Sci 2020; 16(10): 43-49, https://www.researchgate.net/publication/349289409_Effect_of_Benson_Relaxation_and_Aromatherapy_on_Blood_Glucose_Levels_in_Patients_With_Type_II_Diabetes_Mellitus